CLINICAL TRIAL: NCT07166484
Title: Assessment of the Effect of the Product RV2666C Formula LA2984 Compared to an Untreated Area With an Epidermally Ablated Skin Model Obtained With an Erbium YAG Laser on Adults Presenting IV to VI Skin Phototype
Status: Not yet recruiting | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV2666C20250434
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test Group
  Interventions: Other: Cosmetic product RV2666C LA2984

INTERVENTIONS:
Other: Cosmetic product RV2666C LA2984 — The product is applied, according to randomization, on an area located on the anterior side of the forearm, following the laser YAG act, once a day and under occlusion from Day 1 to Day 3 included. Then it is applied twice a day in an open way from Day 4 until Day 18 included.

SUMMARY:
In this study, we assess the efficacy of a cosmetic product in adults with IV to VI skin phototype.

This study is conducted as a monocentric, controlled, compared with an untreated area and randomized for the area of product application.

To perform this clinical study, minimum 20 - maximum 24 subjects (man or woman), aged from 18 to 50 years are enrolled.

The subjects applied the investigational product on an area located on the anterior side of the forearm, following the laser YAG act, once a day and under occlusion from Day 1 to Day 3 included. Then it is applied twice a day in an open way from Day 4 until Day 18 included.

10 visits are planned:

* Visit 1: Inclusion visit = Day 1
* Visit 2 to Visit 5: Intermediate visits = Day 2 to Day 5
* Visit 6: Intermediate visit = Day 8
* Visit 7: Intermediate visit = Day 10
* Visit 8: Intermediate visit = Day 12
* Visit 9: Intermediate visit = Day 15
* Visit 10: End of study visit = Day 19-1

ELIGIBILITY:
Main inclusion criteria :

* Man or woman from 18 to 50 years old
* Phototype IV to VI according to the Fitzpatrick classification
* Subject smoking ≤ 10 cigarettes/day containing nicotine, paper or e-cigarette equivalent
* Subject agreeing not to expose his forearms to UV (natural or artificial) throughout the duration of the study and up to 3 months after the end of participation in the study
* Subject protected by a tetanus vaccination according to the vaccination schedule established by the Public Health Agency

Main non-inclusion criteria:

* Subject suffering from a disease liable to affect the wound healing process according to the opinion of the investigator
* Subject with a known history of allergy or contact dermatitis induced in particular by the latex, the plaster, the local anesthetic, the local antiseptic or one of the components of the study product
* Subject with a disease including skin disease in progress on the upper limbs that may interfere with the interpretation of the evaluation criteria according to the opinion of the investigator
* Topical or oral treatment established or modified during the previous weeks or planned to be established or modified during the study, liable to interfere with the evaluation of the efficacy or cutaneous tolerance of the investigational product according to the investigator's assessment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study is disseminated to the database of potential subjects by email and, if needed, by telephone, describing study title,name(s), address(es) and contacts of the study site(s), name of the Principal Investigator, the parameter(s) in study, study inclusion and exclusion criteria, study objective(s), groups of treatment, namely, if experimental or comparative products are tested, potential risks of adverse events and study duration.
  The subjects that manifested interest in participating in the study might be contacted by telephone.
  Screening questions are asked in order to screen the main inclusion and exclusion criteria Subjects' answers to the telephonic recruitment are evaluated by the Principal Investigator who decides if the subject is to be selected for the recruitment visit.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound healing | Day 1 - Visit 1, Day 2 - Visit 2, Day 3 - Visit 3, Day 4 - Visit 4, Day 5 - Visit 5, Day 8 - Visit 6, Day 10 - Visit 7, Day 12 - Visit 8, Day 15 - Visit 9 and Day 19 - Visit 10.
  The wound disappearance is assessed by the investigator by clinical exam of the skin and from standardized photographs taken with a C Cube Caméra©.
The erythema of the skin | Day 1 - Visit 1 (before and after laser YAG act), Day 2 - Visit 2, Day 3 - Visit 3, Day 4 - Visit 4, Day 5 - Visit 5, Day 8 - Visit 6, Day 10 - Visit 7, Day 12 - Visit 8, Day 15 - Visit 9 and Day 19 - Visit 10.
  The erythema of the skin is assessed objectively using treatment software from standardized photographs using a C Cube Camera©.
The pigmentation of the skin | Day 1 - Visit 1 (before and after laser YAG act), Day 2 - Visit 2, Day 3 - Visit 3, Day 4 - Visit 4, Day 5 - Visit 5, Day 8 - Visit 6, Day 10 - Visit 7, Day 12 - Visit 8, Day 15 - Visit 9 and Day 19 - Visit 10.
  The pigmentation of the skin is assessed objectively using treatment software from standardized photographs using a C Cube Camera©.
The skin marks | Day 2 - Visit 2, Day 3 - Visit 3, Day 4 - Visit 4, Day 5 - Visit 5, Day 8 - Visit 6, Day 10 - Visit 7, Day 12 - Visit 8, Day 15 - Visit 9 and Day 19 - Visit 10.
  The skin marks are evaluated by the investigator at the end of the study using standardized photographs taken with a C Cube© Camera and using an NRS-type evaluation scale from 0 to 10.
The wound healing quality | Day 8 - Visit 6, Day 10 - Visit 7, Day 12 - Visit 8, Day 15 - Visit 9 and Day 19 - Visit 10.
  The wound healing quality is evaluated by the investigator at the end of the study using standardized photographs taken with a C Cube© Camera and using an NRS-type evaluation scale from 0 to 10.
The global efficacy of the product | Day 19 - Visit 10
  The global efficacy of the product is assessed by the subject with a 7-questions questionnaire.
The transepidermal water loss | Day 1 - Visit 1 (before and after laser YAG act), Day 2 - Visit 2, Day 3 - Visit 3, Day 4 - Visit 4, Day 5 - Visit 5, Day 8 - Visit 6, Day 10 - Visit 7, Day 12 - Visit 8, Day 15 - Visit 9 and Day 19 - Visit 10.
  The transepidermal water loss is measured by a clinical research technician using a Vapometer©.
Standardized photographs in an illustrative purpose | Day 1 - Visit 1 (before and after laser YAG act), Day 2 - Visit 2, Day 3 - Visit 3, Day 4 - Visit 4, Day 5 - Visit 5, Day 8 - Visit 6, Day 10 - Visit 7, Day 12 - Visit 8, Day 15 - Visit 9 and Day 19 - Visit 10.
  Photographs in 2D and 3D are taken using a C Cube Camera©.

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Research Center, Toulouse, France, France